CLINICAL TRIAL: NCT00068757
Title: Phase I Study of Lonafarnib (SCH66336) in Combination With Herceptin Plus Paclitaxel in HER 2 NEU Overexpressing Breast Cancer
Brief Title: Lonafarnib, Trastuzumab, and Paclitaxel in Treating Patients With HER2/Neu-Overexpressing Stage IIIB, Stage IIIC, or Stage IV Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: EORTC-16023-10051; EORTC-16023-10051; SPRI-P01900
Record Dates: First submitted 2003-09-10; First posted 2003-09-11 (Estimated); Last update posted 2012-09-12 (Estimated); Status verified 2012-09

CONDITIONS: Breast Cancer
Keywords: recurrent breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; male breast cancer; HER2-positive breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — Trastuzumab; lonafarnib; Paclitaxel

INTERVENTIONS:
Biological: trastuzumab
Drug: lonafarnib
Drug: paclitaxel
Other: pharmacological study

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as paclitaxel, work in different ways to stop tumor cells from dividing so they stop growing or die. Lonafarnib may stop the growth of tumor cells by blocking the enzymes necessary for their growth. Monoclonal antibodies, such as trastuzumab, can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Combining lonafarnib and trastuzumab with paclitaxel may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of lonafarnib when given together with trastuzumab and paclitaxel in treating patients with HER2/neu-overexpressing stage IIIB, stage IIIC, or stage IV breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose and recommended phase II dose of lonafarnib in combination with trastuzumab (Herceptin®) and paclitaxel in patients with HER2/neu-overexpressing stage IIIB, IIIC, or IV breast cancer.
* Determine the qualitative and quantitative toxicity of this regimen in these patients.

Secondary

* Determine the pharmacokinetic profiles of these drugs in these patients.
* Correlate the pharmacodynamics with the pharmacokinetics of this regimen in these patients.
* Correlate the pharmacokinetics and pharmacodynamics of this regimen with observed toxicity in these patients.
* Determine the response to this regimen in patients with measurable disease.

OUTLINE: This is a nonrandomized, open-label, multicenter, dose-escalation study of lonafarnib.

* Course 1: Patients receive a loading dose of trastuzumab (Herceptin®) IV over 90 minutes on day 1 and over 30 minutes on days 8 and 15. Patients also receive paclitaxel IV over 3 hours on day 1.
* Course 2: Patients receive trastuzumab IV over 30 minutes on days 1, 8, and 15 and paclitaxel IV over 3 hours on day 2. Patients also receive oral lonafarnib twice daily on days 3-21.
* Course 3 and all subsequent courses: Patients receive oral lonafarnib twice daily on days 1-21; trastuzumab IV over 30 minutes on days 1, 8, and 15; and paclitaxel IV over 3 hours on day 1.

Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of lonafarnib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed every 8 weeks until disease progression.

PROJECTED ACCRUAL: A total of 3-36 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed breast cancer

  * Stage IIIB, IIIC, or IV
* HER2/neu overexpression

  * 3+ by immunohistochemistry

    * 2+ allowed if positive fluorescent in situ hybridization
* Disease meets the following treatment criteria:

  * Paclitaxel/trastuzumab (Herceptin®) may be appropriate therapy
  * Anthracycline therapy is not a suitable approach
* No clinical signs of CNS involvement
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Male or female

Menopausal status

* Not specified

Performance status

* ECOG 0-2 OR
* WHO 0-2

Life expectancy

* Not specified

Hematopoietic

* Neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10.0 g/dL (6.2 mmol/L)

Hepatic

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase less than 2.5 times ULN (5 times ULN if liver metastases are present)
* AST and ALT less than 2.5 times ULN (5 times ULN if liver metastases are present)

Renal

* Creatinine clearance at least 40 mL/min

Cardiovascular

* Cardiac ejection fraction normal by MUGA
* QTc interval no greater than 440 msec
* No cardiac dysfunction

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for up to 3 months after study participation
* No concurrent severe/unstable systemic disease
* No infection
* No circumstances that would preclude study participation (e.g., alcoholism or substance abuse)
* No psychological, familial, sociological, or geographical condition that would preclude study compliance and follow-up

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 1 year since prior trastuzumab
* No concurrent prophylactic growth factors

Chemotherapy

* More than 1 year since prior paclitaxel
* More than 4 weeks since other prior chemotherapy

Endocrine therapy

* More than 1 day since prior hormonal therapy
* More than 2 days since prior high-dose chronic steroids
* More than 2 days since prior ethinyl estradiol
* No concurrent high-dose chronic steroids
* No concurrent ethinyl estradiol

Radiotherapy

* More than 4 weeks since prior radiotherapy

Surgery

* Not specified

Other

* More than 2 days since prior administration of and no concurrent CYP3A4 inducers or inhibitors, including any of the following:

  * Gestodene
  * Itraconazole
  * Ketoconazole
  * Cimetidine
  * Erythromycin
  * Carbamazepine
  * Phenobarbital
  * Phenytoin
  * Rifampin
  * Sulfinpyrazone
* No concurrent grapefruit juice
* No other concurrent anticancer agents
* No other concurrent investigational therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2003-08; Primary Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity and maximum tolerated dose as measured by CTC v 2.0

SECONDARY OUTCOMES:
Translational research
Pharmacokinetics (PK) and pharmacodynamics (PD)
Clinical response as measured by RECIST criteria

CONTACTS AND LOCATIONS:
Overall Officials: Jan H. M. Schellens, MD, PhD, Study Chair — The Netherlands Cancer Institute
Locations (3):
- Institut Jules Bordet, Brussels, Belgium
- Institut Curie Hopital, Paris, France
- Netherlands Cancer Institute - Antoni van Leeuwenhoek Hospital, Amsterdam, Netherlands